CLINICAL TRIAL: NCT04003532
Title: Evaluation of the Loop-mediated Amplification Assay and Direct-Blood PCR-Nucleic-Acid Lateral Flow Immuno-Assay for the Diagnosis and/or as Test-of-Cure in Patients With Visceral Leishmaniasis in Ethiopia
Brief Title: LAMP Assay for the Diagnosis of Visceral Leishmaniasis
Acronym: EvaLAMP
Status: Completed | Type: Observational
Sponsor: Prof. Dawit Wolday (Other)
Collaborators: European and Developing Countries Clinical Trials Partnership (EDCTP) (Other Government); Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other)
Responsible Party: Sponsor-Investigator, Prof. Dawit Wolday, Associate Professor of Medicine, Mekelle University
Organization: Mekelle University (Other)
Other Study IDs: TMA2016SF-1437
Record Dates: First submitted 2019-06-27; First posted 2019-07-01 (Actual); Last update posted 2023-12-20 (Actual); Status verified 2023-12

CONDITIONS: Visceral Leishmaniasis
Keywords: Diagnosis; Test-of-Cure; HIV co-infection; Loop-mediated amplification assay; PCR; Nucleic-acid Lateral Flow Immunoassay
MeSH Terms: conditions — Leishmaniasis, Visceral; Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Whole-blood
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study will evaluate the of the loop-mediated amplification assay (LAMP) as a diagnostic as well as a Test-of-Cure (ToC) for visceral leishmaniasis (VL) in an endemic area in Ethiopia. Furthermore, we aim to further development of the direct-blood PCR-Nucleic Acid Lateral-Flow Immuno-Assay (dB-PCR-NALFIA) as a novel diagnostic tool for VL and its subsequent evaluation in the field.

DETAILED DESCRIPTION:
Leishmaniasis is among the World's important neglected infectious diseases (NIDs). The WHO estimates that 350 million people are at risk of contracting leishmaniasis. Visceral leishmaniasis (VL) is the most severe form of the disease. Ethiopia has been recently listed by WHO among the fourteen countries in the world with the highest burden of VL. The development of novel point-of-care (PoC) diagnostics and/or a Test-of-Cure (ToC) for VL is deemed a key priority research area. In several endemic areas current gold standard diagnosis and monitoring of treatment efficacy of VL is based on parasite detection or serology. However, these tests are either not available for routine use or lack sufficient sensitivity and specificity, in particular in HIV co-infected patients. Though molecular tests such as PCR have become popular choices as a tool to diagnose VL, monitor treatment response and predict relapse, these techniques require technical skill and equipment and are considerably more expensive. Recent advances in diagnostics has been the development of LAMP with several advantages, such as no need for thermocycler, high specificity, simple read-out and no cold chain requirements. Therefore, LAMP has emerged as a powerful tool for PoC diagnostics. Its clinical utility as PoC diagnosis and/or ToC for VL in the African setting is, however, hardly known.

Here, the investigators will evaluate the utility of the LAMP as a PoC and/or ToC for VL in an endemic area in Ethiopia. The performance of the LAMP assay as a diagnostic tool will be evaluated in newly diagnosed VL cases confirmed by parasite detection and/or PCR. Furthermore, the use of the assay as ToC will be determined by evaluating the performance of the assay in VL patients confirmed cured at day 17 of therapy, as assessed by negative parasite and/or PCR results. Additionally, the investigators plan to utilize a newly developed rapid molecular platform, db-PCR-NALFIA, which does not require DNA extraction, has an internal amplification control and simple read-out. The investigators will evaluate the utility of both assays also in patients co-infected with HIV. The results may have major policy implications as the application represents a concept that could enhance evidence- based translation of research to improve public health practice by contributing to leishmaniasis management guidelines - with overarching impacts for National, Regional and Global programs.

ELIGIBILITY:
Inclusion Criteria:

* Clinical evidence consistent with VL confirmed by microscopy (+ culture) and/or PCR

Exclusion Criteria:

* Treatment with any anti-leishmanial drugs within the previous 3 months
* Not capable of understanding or complying with the study protocol
* Refusal to consent and participate in to the study

Ages: 5 Years to 90 Years | Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: VL suspected cases will be recruited from Ayder Referral Hospital, Mekelle University College of Health Sciences - (MUCHS) in Mekelle City, the capital of Tigray Regional State in Northern Ethiopia, where VL is highly endemic in the area. Patients seeking care at the hospital will be eligible and screened for inclusion in the study.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Actual)
Dates: Start 2018-10-01 (Actual); Primary Completion 2022-06-30 (Actual); Study Completion 2023-06-30 (Actual)

PRIMARY OUTCOMES:
Number of participants correctly diagnosed with VL as assessed by LAMP assay | Baseline
  Performance of the LAMP will be compared to gold- standard diagnostic procedures, including parasite detection and/or PCR-technology
Number of participants treated for VL and identified as cured (ToC) at day 17 post-treatment based on the assessment by LAMP assay | Baseline
  LAMP will be compared to gold- standard diagnostic procedures, including parasite detection and/or PCR-technology

SECONDARY OUTCOMES:
Number of participants co-infected with HIV correctly diagnosed with VL as well as treated participants identified as cured (ToC) at day 17 based on the assessment by LAMP assay | 17 days
  LAMP will be compared to gold-standard diagnostic procedures, including parasite detection and/or PCR-technology
Number of participants correctly diagnosed as VL based on db-PCR-NALFIA technology | Baseline
  The investigators will develop db-PCR-NALFIA technology for the diagnosis of VL, i.e. sample preparation and result read-out will be adopted using db-PCR-NALFIA technology as PoC platform. It's performance will be evaluated against gold-standard.

CONTACTS AND LOCATIONS:
Overall Officials: Amanuel Haile, MD, Study Chair — Mekelle University College of Health Sciences
Locations (1):
- Mekelle University College of Health Sciences, Mek'ele, Ethiopia

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual patient data for all primary and secondary outcome measures will be made available to anyone who submit requests.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: After 12 months of completion of project
Access Criteria: Data access requests will be first reviewed by the project's steering committee to ensure that all requested analyses can be achieved with the available study data.

REFERENCES:
- [Result] Hagos DG, Schallig HDFH, Kiros YK, Abdulkadir M, Wolday D. Performance of rapid rk39 tests for the diagnosis of visceral leishmaniasis in Ethiopia: a systematic review and meta-analysis. BMC Infect Dis. 2021 Nov 17;21(1):1166. doi: 10.1186/s12879-021-06826-w. PMID 34789175
- [Result] Hagos DG, Kiros YK, Abdulkader M, Arefaine ZG, Nigus E, Schallig HHDF, Wolday D. Utility of the Loop-Mediated Isothermal Amplification Assay for the Diagnosis of Visceral Leishmaniasis from Blood Samples in Ethiopia. Am J Trop Med Hyg. 2021 Jul 26;105(4):1050-1055. doi: 10.4269/ajtmh.21-0334. PMID 34310340
- [Result] Hagos DG, Kebede Y, Abdulkader M, Nigus E, Gessesse Arefaine Z, Nega G, Schallig HDF, Wolday D. Effect of rK39 testing in guiding treatment initiation and outcome in patients with visceral leishmaniasis in Ethiopia: A prospective cohort study. PLoS One. 2021 Jun 14;16(6):e0253303. doi: 10.1371/journal.pone.0253303. eCollection 2021. PMID 34125865